CLINICAL TRIAL: NCT03831568
Title: Prevalence and Use of Mechanical Cough Augmentation in Children With Neuromuscular Disorders in Norway
Brief Title: Mechanical Cough Augmentation in Children With NMD
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital of North Norway (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); Sorlandet Hospital HF (Other Government)
Responsible Party: Principal Investigator, Brit Hov, Physiotherapist, MSc, Oslo University Hospital
Other Study IDs: MIE 2016_14321; 17/9232 (Registry Identifier: NPR); Hov_2017 (Registry Identifier: NR LTMV)
Record Dates: First submitted 2017-11-27; First posted 2019-02-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Neuromuscular Diseases; Children, Only; Airway Clearance Impairment; Cough
Keywords: Airway management; Cough; Neuromuscular diseases; Pediatrics; Mechanical insufflation-exsufflation
MeSH Terms: conditions — Neuromuscular Diseases; Cough

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with given device for mechanical cough

SUMMARY:
The study investigates the prevalence and use of mechanical insufflation - exsufflation (MI-E) in children with Neuromuscular disorders (NMD) in Norway. The NMD related prevalence of MIE use in Norway will be described and possible regional differences regarding use will be assessed.

DETAILED DESCRIPTION:
Neuromuscular diseases (NMD) in children are severe, possibly life-threatening orphan conditions. Respiratory tract infections and lung complications are the main causes of increased morbidity and mortality.

The use of mechanical cough augmentation with insufflation-exsufflation (MIE) is a strategy to treat and prevent. Possible major benefits are described, but optimal settings for best efficacy and comfort in children are not established.

The main objective is to determine the prevalence and use of MIE among children with NMD in Norway. All children with NMD < 18 years which has received a machine for MI-E will be invited to participate in the study.

The participants will be asked to complete two questionnaires. In addition will information from the data card in the MI-E machines give information about use. The information will be linked to the National register for Long term mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria: ,

* Received a MI-E device
* Neuromuscular disease
* < 18 years

Exclusion Criteria:

- None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with neuromuscular disorder bellow 18 years that has received a machine for MI-E.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Residency | At one point (1 day)
  Name of county
Indication for use | At one point (1 day)
  Prevention or treatment purposes from questionnaire
Diagnosis | 01.01.2018
  International Classification of Diseases - 10 diagnosis

SECONDARY OUTCOMES:
Health related quality of life | One time at completion of questionaire
  The DISABKIDS Chronic Generic Module (DCGM-37) is a questionnaire measuring general health-related quality of life (HRQoL) and the level of distress caused by a chronic disease at 3 domains (mental, social and physical) in 6 dimensions: Independence, Emotion, Social inclusion, Social exclusion, Limitation and Treatment. Each item is scored on a five-point Likert scale which indicates behavior or feelings as 1 = never, 2 = seldom, 3 = quite often, 4 = very often and 5 = always. There is one form to be filled in by children 8 to 18 years of age, and one form by their parents. The sum of scores within each dimension makes up the raw score, which is transformed linearly into a score ranging from 0 to 100. The scores are added and further transformed into a total HRQOL score with a range 0 to 100 with higher scores indicating higher HRQOL.
Settings in use | One time at completion of questionaire
  Recorded from data card in MIE machine
Opinion on treatment | One time at completion of questionaire
  A purpose made questionnaire including questions with predefined categorical data in no order, and 2 questions using a Visual Analog Scale 0-10 to score perceived benefit of the treatment where 0 indicates not important at all and 10 indicates very important.

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Hovland, PhD, Principal Investigator — MD
Locations (1):
- Oslo university hospital, Oslo, Norway